CLINICAL TRIAL: NCT06818604
Title: Comparison Between CPAP and BiPAP for Management of Sleep Disordered Breathing in Cervical Spinal Cord Injury Patients: a Pilot Randomized Controlled Study
Brief Title: Comparing CPAP and BiPAP for Sleep-Disordered Breathing in People with Cervical Spinal Cord Injuries
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Najib Ayas, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H24-01212
Record Dates: First submitted 2025-01-13; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2024-12

CONDITIONS: Spinal Cord Injuries (SCI); Sleep Disordered Breathing (SDB); Sleep Apnea; Cervical Spinal Cord Injruy
Keywords: sleep disordered breathing; Cervical Vertebrae; Obstructive Sleep Apnea; Spinal Cord Injuries; Positive Pressure Respiration; Continuous Positive Airway Pressure; Sleep Quality; Quadriplegia; Polysomnography; Tetraplegia; Sleep Wake Disorders; Diaphragmatic Paralysis; Autonomic Dysreflexia; Muscle Weakness; Nocturnal Hypoventilation; Phrenic Nerve; Pulmonary Atelectasis; Spinal Cord Compression; Ventilator Weaning; Neurological Rehabilitation; Sleep Disorders; Activities of Daily Living
MeSH Terms: conditions — Spinal Cord Injuries; Sleep Apnea Syndromes; Sleep Apnea, Obstructive; Sleep Initiation and Maintenance Disorders; Quadriplegia; Sleep Wake Disorders; Respiratory Paralysis; Autonomic Dysreflexia; Muscle Weakness; Pulmonary Atelectasis; Spinal Cord Compression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CPAP Therapy (Experimental)
  Interventions: Device: CPAP
- BiPAP Therapy (Experimental)
  Interventions: Device: BiPAP

INTERVENTIONS:
Device: CPAP — Participants randomized to this group will receive auto-CPAP therapy. The device will be initiated by a respiratory therapist at GF Strong Rehabilitation Centre. Settings will be adjusted to achieve a device efficacy index < 5 events per hour.
  Arms: CPAP Therapy
Device: BiPAP — Participants will receive BiPAP S mode therapy for 4 weeks. The device will be initiated by a respiratory therapist at GF Strong Rehabilitation Centre with initial settings of IPAP 8 cmH2O and EPAP 3 cmH2O. Settings will be modified to a maximum tolerated level to achieve a tidal volume of 8 mL/kg ideal body weight and SpO2 > 95%. Overnight oximetry will be performed to ensure at least 4 hours of device use, and settings will be adjusted to achieve a DEI < 5 events per hour.
  Arms: BiPAP Therapy

SUMMARY:
Sleep-disordered breathing (SDB) is common in individuals with cervical spinal cord injuries, with studies suggesting prevalence rates ranging from 27% to 62%. The condition often leads to daytime sleepiness, fatigue, and poor participation in rehabilitation. Positive airway pressure therapy can be used to treat the condition; however, some individuals find continuous positive airway pressure (CPAP), which applies the same pressure during inhalation and exhalation, difficult to use. Bilevel positive airway pressure (BiPAP) offers different pressures for inhalation and exhalation, which may be more comfortable and potentially improve adherence in this patient population. However, limited evidence compares CPAP and BiPAP in individuals with cervical spinal cord injuries.

This pilot study will enroll 32 adult participants with cervical spinal cord injuries who have moderate to severe SDB (defined as an AHI of 15 events/hour or greater). Participants will be randomly assigned to either CPAP or BiPAP therapy for 4 weeks. Device usage per night will be measured, and data on daytime sleepiness, fatigue, and sleep quality will be collected at baseline, 2 weeks, and 4 weeks. The investigators aim to determine whether BiPAP improves adherence and symptoms compared to CPAP in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 19 years
* Cervical spinal cord injury (ASIA A, B, or C). This will include patients with upper (C1-C4) and lower (C5-C7) spinal cord injuries
* Presence of sleep disordered breathing, defined as AHI > =15 events/hour by home sleep apnea test (HSAT)

Exclusion Criteria:

* On CPAP or BiPAP prior to spinal cord injury
* Hypoventilation syndrome (elevated venous carbon dioxide, PvCO2>50 mm Hg)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Adherence to PAP Therapy | 4 weeks
  Median hours of PAP device use per night, objectively measured via device download. Additional metrics include: % days used >4 hrs/night, total # of days used, total # of hours used.

SECONDARY OUTCOMES:
Daytime Sleepiness | 4 weeks
  Measured using the Epworth Sleepiness Scale (ESS). ESS is a self-administered questionnaire that asks participants to rate their likelihood of dozing off or falling asleep in eight different situations that are common in daily life. Scores range from 0 to 24, with higher scores indicating greater daytime sleepiness.
Sleep Quality | 4 weeks
  Measured using the Pittsburgh Sleep Quality Index (PSQI). The PSQI is a self-rated questionnaire that assesses sleep quality over the past month. The PSQI yields seven component scores, each ranging from 0 to 3, which are summed to produce a global PSQI score ranging from 0 to 21. Higher global PSQI scores indicate poorer sleep quality.
Fatigue | 4 weeks
  Measured using the PROMIS-Fatigue (PROMIS-F) scale. The PROMIS-F is a standardized, self-reported measure of fatigue. PROMIS-F T-scores are standardized to a mean of 50 and a standard deviation of 10. Higher T-scores indicate greater fatigue.
PAP side effects | 4 weeks
  Assessed using a PAP therapy side effect survey. This survey will collect information about any side effects experienced by participants as a result of using the PAP devices.
Recruitment Rate | 4 weeks
  Helps assess the feasibility of recruiting this specific patient population for future, larger studies. Also helps us understand if there are any barriers to participation that need to be addressed in future research. Recruitment rate will be assessed as the average number of participants enrolled per month during the recruitment period.

CONTACTS AND LOCATIONS:
Locations (1):
- GF Strong Rehabilitation Centre, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No